CLINICAL TRIAL: NCT01987089
Title: The Efficacy of CBT-I in Alcoholics & Its Effects on Remission & Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Pennsylvania (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NURA-017-13S; 1IK2CX000855 (NIH); 01468 (Other: Philadelphia Veterans Affairs Medical Center)
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Insomnia
Keywords: Insomnia; Sleep initiation and maintenance disorder; Alcoholism; Cognitive behavioral therapy for insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Alcoholism | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT-I (Experimental): Eight Session CBT-I: Cognitive Behavioral therapy is conducted in 8 individual sessions with the study clinician. Session 1 serves as an orientation. No active treatment is delivered at this time. Sessions 2 & 3 are used to deliver the three main components of the intervention which are Sleep Restriction (SRT), Stimulus Control, and Sleep Hygiene. All but two of the remaining sessions are dedicated to the titration of total sleep time and to ensuring patient adherence. One session (session 5) entails the delivery of a specific form of cognitive therapy. The final session (session 8) is used to engage in a relapse-prevention didactic, i.e., to review first, how insomnia becomes chronic and second, the strategies that are likely to abort an extended episode of insomnia.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
- QDT (Placebo Comparator): This form of placebo therapy has been commonly used in prior studies investigating behavioral interventions for insomnia. The therapist presents the QDT as a means to eliminate "conditioned arousal," occurring after nocturnal arousal using 8 sessions on a weekly basis. The therapist initially helps the subject to develop a chronological 12-item hierarchy of commonly practiced activities on awakening at night, like opening eyes and clock watching. As a next step, the subject develops 6 imaginable scenes of himself/herself engaged in neutral activities like reading a newspaper. The therapist then helps the subject pair the neutral scenes with the items from the 12-item hierarchy, which is then practiced by the subject 2 hours before bedtime.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — Eight Session CBT-I: Cognitive Behavioral therapy is conducted in 8 individual sessions with the study clinician.

SUMMARY:
Insomnia is a highly prevalent disorder in those recovering from alcoholism. It has been associated with anxiety and depressive symptoms, as well as an increased risk of relapse back to the drinking.

Cognitive Behavioral Therapy for Insomnia (CBT-I), a non-pharmacologic approach is the recommended standard of care for insomnia. Some preliminary studies have shown that CBT-I may be efficacious for insomnia during recovery.

The current study proposes to use a standard 8-week CBT-I to treat the insomnia with a post-treatment follow-up at 3- and 6-months (after treatment). Further, it will evaluate if an improvement in the insomnia is associated with an improvement in the underling alcoholism and the daytime functioning. On an exploratory basis, the association of a first-degree family history of alcoholism with the insomnia severity and treatment response will also be evaluated.

DETAILED DESCRIPTION:
Eligible subjects will be Veterans with alcohol dependence during their first year of recovery, 21-65 years old, with ISI total score of 15 or more, medically and psychiatrically stable, and without dependence on other drugs (with the exception of nicotine and marijuana).

The proposed study will consist of a single-blind trial comparing CBT-I against a behavioral placebo intervention (Quasi-Desensitization Therapy, QDT).

Baseline assessments conducted over a month will comprehensively evaluate for the addiction, psychiatric, sleep and medical disorders, as well as for a family history of alcohol dependence.

Once the subject is seen to be eligible for the study he will be randomized to either the CBT-I or the QDT arm, and treated for the next weeks. The primary outcome measure for insomnia will be the Insomnia Severity Index. The primary outcome measure for alcohol dependence will be the percent days abstinent (on the Time Line Follow Back measure, TLFB), and the daytime symptoms will be assessed using the Short Form-12 item scale (SF-12, for self reported well-being), the Beck Depression Inventory (BDI, for depressive symptoms), and the State Trait Anxiety Inventory (STAI, for anxiety symptoms).

After completion of the treatment phase, subjects will be followed up 3 months and 6 months later, to assess for changes over time in their insomnia, alcohol use, and daytime functioning.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Veterans between the ages of 21 and 70 years
* DSM IV diagnosis of alcohol dependence over the past year (as determined by the Structured Clinical Interview for DSM-IV Axis I Disorders [SCID-I])
* Self-reported sleep latency or wake time after sleep onset >30 min on three or more nights per week for 1 month and a score of 15 or more on the Insomnia Severity Index (ISI)
* No current alcohol withdrawal symptoms at baseline: CIWA score < 8 (CIWA is the Clinical Institute Withdrawal Assessment scale for alcohol withdrawal signs and symptoms)
* Abstain for at least 4 weeks from heavy drinking, and < 12 months of abstinence from heavy drinking prior to the baseline study assessments, as assessed by subjective report or breathalyzer
* Ability to speak, understand and print in English
* Capacity to give written informed consent

Exclusion Criteria:

* DSM-IV criteria for dependence on any other substance including benzodiazepines (and excluding nicotine dependence)
* Positive urine drug screen for opioids, cocaine, or amphetamine (positive screen for Tetra Hydro Cannabinol is not considered an exclusion criteria)
* Patient is currently in alcohol withdrawal as assessed by the Clinical Institute Withdrawal Assessment Scale (CIWA) total score of 8 or more
* A lifetime DSM-IV diagnosis of Bipolar I or II disorder, Schizophrenia, or other psychotic disorder, as determined on the SCID-I, and current (past month) DSM-IV diagnosis of Major Depressive Disorder
* Presence of unstable medical diagnosis e.g. congestive heart failure, leading to interference with sleep, as reported on history, examination, and/or review of clinical chart during baseline assessments
* Current use of any medications that may influence the drinking behavior, e.g. naltrexone or acamprosate
* Evidence of severe cognitive impairment as assessed by the Blessed Orientation-Memory-Concentration (BOMC) test weighted score
* Untreated patients with the diagnosis of moderate-severe obstructive sleep apnea with Total Apnea-Hypopnea Index (AHI-T) of 15 events/hour of sleep
* Subject's inability to give informed consent

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-08-15 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Subhajit Chakravorty, MD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 83 was the anticipated recruitment target sample and our final recruitment sample was 63
Groups:
- Cognitive Behavioral Therapy for Insomnia (CBT-I): Eight Session CBT-I: Cognitive Behavioral therapy is conducted in 8 individual sessions with the study clinician. Session 1 serves as an orientation. No active treatment is delivered at this time. Sessions 2 & 3 are used to deliver the three main components of the intervention which are Sleep Restriction (SRT), Stimulus Control, and Sleep Hygiene. All but two of the remaining sessions are dedicated to the titration of total sleep time and to ensuring patient adherence. One session (session 5) entails the delivery of a specific form of cognitive therapy. The final session (session 8) is used to engage in a relapse-prevention didactic, i.e., to review first, how insomnia becomes chronic and second, the strategies that are likely to abort an extended episode of insomnia.
  Cognitive Behavioral Therapy for Insomnia (CBT-I): Eight Session CBT-I: Cognitive Behavioral therapy is conducted in 8 individual sessions with the study clinician.
- Quasi Desensitization Therapy (QDT): This form of placebo therapy has been commonly used in prior studies investigating behavioral interventions for insomnia. The therapist presents the QDT as a means to eliminate "conditioned arousal," occurring after nocturnal arousal using 8 sessions on a weekly basis. The therapist initially helps the subject to develop a chronological 12-item hierarchy of commonly practiced activities on awakening at night, like opening eyes and clock watching. As a next step, the subject develops 6 imaginable scenes of himself/herself engaged in neutral activities like reading a newspaper. The therapist then helps the subject pair the neutral scenes with the items from the 12-item hierarchy, which is then practiced by the subject 2 hours before bedtime.
  Cognitive Behavioral Therapy for Insomnia (CBT-I): Eight Session CBT-I: Cognitive Behavioral therapy is conducted in 8 individual sessions with the study clinician.
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy for Insomnia (CBT-I) | Quasi Desensitization Therapy (QDT)
Started | 31 | 32
Completed | 30 | 28
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Cognitive Behavioral Therapy for Insomnia: Eight Session CBT-I: Cognitive Behavioral therapy is conducted in 8 individual sessions with the study clinician. Session 1 serves as an orientation. No active treatment is delivered at this time. Sessions 2 & 3 are used to deliver the three main components of the intervention which are Sleep Restriction (SRT), Stimulus Control, and Sleep Hygiene. All but two of the remaining sessions are dedicated to the titration of total sleep time and to ensuring patient adherence. One session (session 5) entails the delivery of a specific form of cognitive therapy. The final session (session 8) is used to engage in a relapse-prevention didactic, i.e., to review first, how insomnia becomes chronic and second, the strategies that are likely to abort an extended episode of insomnia.
  Cognitive Behavioral Therapy for Insomnia (CBT-I): Eight Session CBT-I: Cognitive Behavioral therapy is conducted in 8 individual sessions with the study clinician.
- Quasi Desensitization Therapy: This form of placebo therapy has been commonly used in prior studies investigating behavioral interventions for insomnia. The therapist presents the QDT as a means to eliminate "conditioned arousal," occurring after nocturnal arousal using 8 sessions on a weekly basis. The therapist initially helps the subject to develop a chronological 12-item hierarchy of commonly practiced activities on awakening at night, like opening eyes and clock watching. As a next step, the subject develops 6 imaginable scenes of himself/herself engaged in neutral activities like reading a newspaper. The therapist then helps the subject pair the neutral scenes with the items from the 12-item hierarchy, which is then practiced by the subject 2 hours before bedtime.
  Cognitive Behavioral Therapy for Insomnia (CBT-I): Eight Session CBT-I: Cognitive Behavioral therapy is conducted in 8 individual sessions with the study clinician.
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy for Insomnia | Quasi Desensitization Therapy | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (10.9) | 51.5 (8.2) | 51.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 28 | 30 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 23 | 29 | 52
  Caucasian | 8 | 3 | 11
  Hispanic | 1 | 1 | 2
Insomnia Severity Index total score (ISI) [Mean (Standard Deviation); unit: units on a scale] — 7-item (0-4 Likert scales) measure yields a total score of 28. The norms for the scale are as follows: 0-7 represents no clinically significant insomnia; 8-14 represents sub threshold insomnia; 15-21 represents clinical insomnia (moderate severity); 21-28 represents clinical insomnia (severe)
  units on a scale | 19.7 (3.5) | 19.0 (3.7) | 19.3 (3.6)
Sleep Onset Latency (SOL, sleep diary) [Mean (Standard Deviation); unit: minutes] | 51.6 (41.4) | 49.3 (34.0) | 50.5 (37.7)
Wake After Sleep Onset (WASO, sleep diary) [Mean (Standard Deviation); unit: minutes] | 44.6 (30.0) | 28.6 (25.5) | 36.7 (28.8)
Total Sleep Time (TST, sleep diary) [Mean (Standard Deviation); unit: minutes] | 317.0 (90.8) | 345.1 (99.5) | 330.8 (95.5)
Percent Days Abstinent (PDA, last 90 days, at screening) [Mean (Standard Deviation); unit: Percent of Days Abstinent] | 38.3 (36.0) | 26.9 (29.2) | 32.5 (32.9)
Drinks per day (DrPDay, last 90 days, at screening) [Mean (Standard Deviation); unit: Number of Drinks Per Day] | 9.1 (9.2) | 8.8 (7.1) | 8.9 (8.1)
Penn Alcohol Craving Scale total score (PACS) [Mean (Standard Deviation); unit: units on a scale] — The PACS is a 5-item scale that evaluates alcohol craving over the last seven days. Item scores range from 0-6 and a total PACS score ranging from 0-30. A higher value on the PACS total score represents an increasing severity of alcohol craving.
  units on a scale | 10.8 (7.5) | 8.2 (7.0) | 9.5 (7.3)
Days Abstinent from Alcohol before Treatment (Abs) [Mean (Standard Deviation); unit: Number of Days] | 86.8 (103.3) | 142.6 (111.6) | 115.2 (110.4)
Physical Composite Score (PCS, SF-12 scale) [Mean (Standard Deviation); unit: units on a scale] — The Physical Composite Scale (PCS) is a scale generated from the 12-item short-form (SF-12) measure. The PCS evaluates the self-reported physical well-being of an individual. The PCS has a range from 0-100, where 0 indicates the lowest level and 100 indicates the highest level of physical health.
  units on a scale | 42.7 (4.6) | 40.4 (5.3) | 41.7 (5.0)
Mental Composite Score (MCS, SF-12 scale) [Mean (Standard Deviation); unit: units on a scale] — The Mental Composite Scale (MCS) is another scale generated from the 12-item short-form (SF-12) measure. The MCS evaluates the self-reported emotional well-being of an individual. The MCS also has a range from 0-100, where 0 indicates the lowest level and 100 indicates the highest level of mental health.
  units on a scale | 44.4 (7.5) | 43.1 (6.4) | 43.9 (6.9)
Beck Depression Inventory total score [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory (BDI) is a 21-item self-reported measure of depressive symptoms, and a recommended measure of next day functioning in studies evaluating insomnia disorder. The BDI generates a total score within a range from 0-63, with higher scores representing increasing severity of depressive symptoms.
  units on a scale | 19.7 (12.4) | 17.2 (10.7) | 18.5 (11.6)
State Trait Anxiety Inventory - trait subscale (STAI-trait) [Mean (Standard Deviation); unit: units on a scale] — The State-Trait Anxiety Inventory (STAI) is a 40-item self-reported measure of state and trait anxiety symptoms. The trait subscale is a recommended measure of next day functioning in studies evaluating insomnia disorder. The STAI trait subscale generates a total score within a range from 20-80, with higher scores representing greater anxiety.
  units on a scale | 45.0 (5.9) | 46.3 (6.0) | 45.6 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insomnia Severity Index - Total Score
Description: Insomnia Severity Index (ISI): This 7-item (0-4 Likert scales) measure yields a total score of 28. The norms for the scale are as follows: 0-7 represents no clinically significant insomnia; 8-14 represents sub threshold insomnia; 15-21 represents clinical insomnia (moderate severity); 21-28 represents clinical insomnia (severe). The scale provides a measure of severity of insomnia (overall), a measure of insomnia subtype, a measure of the diurnal effects of insomnia, and a measure of sleep "satisfaction". The ISI will be completed at baseline and for all the subsequent study-related visits.
Time Frame: 8 weeks, 3 months post-treatment, and 6 months post-treatment
Population: All subjects randomized into either treatment arm and received had 1 or more treatment sessions.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy for Insomnia (CBT-I) | Quasi Desensitization Therapy (QDT)
Number analyzed (Participants) | 31 | 32
units on a scale
  Change at week 8 (Vs baseline) | -10.71 [-13.07 to -8.10] | -8.84 [-10.82 to -6.84]
  Change at 3 mo post-treatment F/U (Vs baseline) | -8.51 [-11.21 to -5.78] | -9.30 [-11.43 to -7.26]
  Change at 6 mo post-treatment F/U (Vs baseline) | -6.89 [-9.48 to -4.29] | -7.29 [-9.50 to -4.63]

2. Primary Outcome: Change in Percent Days Abstinent (PDA) on the Time Line Follow Back Measure
Description: Time Line Follow Back measure (TLFB): The TLFB provides assessment of drinking using a calendar format for the number of standard alcoholic beverages consumed per day. A standard drink, as defined by the National Institutes of Health, is 12 oz of regular beer, 5 oz of regular wine, or 1.5 oz of distilled spirits (e.g. whiskey). Numerous indices may be derived from the TLFB, such as the Percent Days Abstinent (PDA) proposed in this study. The PDA is derived as the percentage of days an individual reports being abstinent from alcohol within a given assessment time period.
Time Frame: 8 weeks, 3 months post-treatment and 6-months post-treatment
Population: All subjects randomized into either treatment arm and received had 1 or more treatment sessions.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of abstinent days
Arm/Group | Cognitive Behavioral Therapy for Insomnia (CBT-I) | Quasi Desensitization Therapy (QDT)
Number analyzed (Participants) | 31 | 32
percentage of abstinent days
  Change at week 8 (Vs baseline) | 0.56 [0.44 to 0.68] | 0.67 [0.55 to 0.80]
  Change at 3 mo post-treatment F/U (Vs baseline) | 0.51 [0.38 to 0.63] | 0.61 [0.50 to 0.74]
  Change at 6 mo post-treatment F/U (Vs baseline) | 0.48 [0.36 to 0.60] | 0.62 [0.50 to 0.74]

3. Other Pre Specified Outcome: Change in PCS From the Short Form - 12 Item (SF-12) Measure
Description: The Physical Component Summary (PCS) scale has a range from 0 (indicating the lowest level of health) to 100 (indicating the best level of health).
Time Frame: 8 weeks, 3 months post-treatment, and 6 months post-treatment
Population: All subjects randomized into either treatment arm and received had 1 or more treatment sessions.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy for Insomnia (CBT-I) | Quasi Desensitization Therapy (QDT)
Number analyzed (Participants) | 31 | 32
units on a scale
  Change at week 8 (Vs baseline) | -1.00 [-3.29 to 1.30] | 0.48 [-2.70 to 3.80]
  Change at 3 mo post-treatment F/U (Vs baseline) | -1.69 [-5.13 to 1.59] | 0.54 [-2.21 to 3.13]
  Change at 6 mo post-treatment F/U (Vs baseline) | -1.18 [-3.10 to 1.00] | -0.25 [-3.41 to 3.18]

4. Other Pre Specified Outcome: Change in MCS From the Short Form - 12 Item (SF-12) Measure
Description: The Mental Component Summary (MCS) scale has a range from 0 (indicating the lowest level of health) to 100 (indicating the best level of health).
Time Frame: 8 weeks, 3 months post-treatment, and 6 months post-treatment
Population: All subjects randomized into either treatment arm and received had 1 or more treatment sessions.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy for Insomnia (CBT-I) | Quasi Desensitization Therapy (QDT)
Number analyzed (Participants) | 31 | 32
units on a scale
  Change at week 8 (Vs baseline) | -3.06 [-8.04 to 1.71] | -1.90 [-5.92 to 2.16]
  Change at 3 mo post-treatment F/U (Vs baseline) | -2.60 [-7.83 to 2.42] | 1.12 [-2.80 to 5.02]
  Change at 6 mo post-treatment F/U (Vs baseline) | -2.07 [-5.90 to 1.64] | 0.89 [-4.32 to 5.84]

ADVERSE EVENTS:
Time Frame: 9 months
Description: This a behavioral treatment intervention study.
Arm/Group | Cognitive Behavioral Therapy for Insomnia (CBT-I) | Quasi Desensitization Therapy (QDT)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 7/31 | 3/32
Other Adverse Events (participants affected / at risk) | 0/31 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cognitive Behavioral Therapy for Insomnia (CBT-I) (N=31) | Quasi Desensitization Therapy (QDT) (N=32)
Cerebrovascular Accident (CVA) (Nervous system disorders) | 0 | 1
Alcohol detoxification (Nervous system disorders) | 4 | 2 — Relapse to drinking
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Residential Psychiatric Treatment (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT01987089/Prot_SAP_000.pdf